CLINICAL TRIAL: NCT04198220
Title: BIO|STREAM.ICM Obesity, Submodule of the BIO|STREAM.ICM Registry
Brief Title: BIO|STREAM.ICM Obesity
Status: Completed | Type: Observational
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: HS064
Record Dates: First submitted 2019-12-12; First posted 2019-12-13 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2020-12

CONDITIONS: Tachycardia Atrial; Atrial Fibrillation; Syncope; Bradycardia; Cryptogenic Stroke
Keywords: Obesity; BIOMONITOR; BIOMONITOR III; Syncope; Cryptogenic stroke; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation; Syncope; Bradycardia; Ischemic Stroke; Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the submodule study is to assess whether a high BMI may influence the sensing performance and the sECG quality of the BIOMONITOR.

DETAILED DESCRIPTION:
This submodule of the BIO|STREAM.ICM registry specifically investigates the performance of the BIOMONITOR in a subset of obese patients with a BMI >30 kg/m2 in order to exclude any concerns regarding impaired ICM sensing performance. These concerns are founded in the increased distance between heart and device electrodes due to fat layers that may attenuate signal detection and therefore sensing performances of the ICM.

ELIGIBILITY:
Inclusion Criteria:

* Patient is already enrolled in the BIO|STREAM.ICM registry
* Patient BMI > 30

Exclusion Criteria:

* Patient clinically indicated for or already implanted with another cardiac active device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population consists of obese patients (BMI > 30 kg/m2) with an implantable cardiac monitor
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
R-wave amplitude | 3 month
  R-wave amplitude at 3-month Home Monitoring observation in patients with a BMI > 30

SECONDARY OUTCOMES:
Amount of 'noise burden' | 3 month
  Measurement of amount of 'noise burden' during the study period
P-wave visibility | 1 month and 3 month
  Measurement of the P-wave visibility at 1- and 3-month Home Monitoring observation

OTHER OUTCOMES:
Incidence of arrhythmias | 3 month
  Assessment of the incidence of arrhythmias in obese patients implanted with an ICM

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Bisignani, Dr., Principal Investigator — Ospedale Civile Ferrari
Locations (1):
- Ospedale Civile Ferrari, Castrovillari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bisignani G, De Bonis S, Pierre B, Lau DH, Hofer D, Sanfins VM, Hain A, Cabanas P, Martens E, Berruezo A, Eschalier R, Milliez P, Lusebrink U, Mansourati J, Papaioannou G, Giacopelli D, Gargaro A, Ploux S. Insertable cardiac monitor with a long sensing vector: Impact of obesity on sensing quality and safety. Front Cardiovasc Med. 2023 Mar 21;10:1148052. doi: 10.3389/fcvm.2023.1148052. eCollection 2023. PMID 37025684